CLINICAL TRIAL: NCT03843177
Title: Association of Ingrown Toenails With Flat Foot, Hallux Abducto Valgus and Hallux Limitus
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Him Shun KEI, MSc Student, Chinese University of Hong Kong
Other Study IDs: 2017.637
Record Dates: First submitted 2019-02-13; First posted 2019-02-15 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Ingrown Toe Nail; Flat Foot; Hallux Abductovalgus; Hallux Limitus
MeSH Terms: conditions — Nails, Ingrown; Flatfoot; Hallux Valgus; Hallux Limitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ingrown toenails
  Interventions: Other: No intervention
- Control

INTERVENTIONS:
Other: No intervention — No intervention will be performed. Only assessment will be done.
  Groups: Ingrown toenails

SUMMARY:
This study will have implications for any healthcare professionals who routinely manage ingrown toenails. Although different conservative and surgical treatment have been suggested, the recurrent rate is still high ranging from 20% to 30%. The objective of this study was to investigate the association of ingrown toenail (IGTN) with flat foot, hallux abducto valgus (HAV) and hallux limitus (HL), and to provide directions for addressing biomechanical risk factors in the prevention of recurrent ingrown toenails. This was the first study to investigate the association of IGTN with flat foot, and the first study in Chinese community to investigate the association of IGTN with HAV or HL.

Participants with ingrown toenails (IGTN) were recruited to this study and compared with control participants with no history of ingrown toenails.

The inclusion criteria for the IGTN group were: (1) history of ingrown toenails on hallux within 1 year and (2) dorso-plantar standing view of foot x-ray taken or to be taken.

The exclusion criteria for the IGTN group were: (1) paediatrics (Age<18), (2) pincer nails / fungal nails, (3) prior existence of osteoarticular surgery in the foot, (4) severe trauma that changes foot morphology, (5) uncontrolled systemic disease, (6) pre-existing neurological diseases and (7) lower limb paralysis or paresis.

The inclusion criterion for the control group was dorso-plantar standing view of foot x-ray taken or to be taken.

The exclusion criteria for the control group were: (1) all the exclusion criteria of IGTN group, (2) history of IGTN in his or her lifetime and (3) flatfoot / first metatarsophalangeal joint pathology as the chief complaint.

The symptomatic foot (or the more symptomatic foot in the case of bilateral involvement) in the IGTN group was examined. The left or right foot of the control group was randomly selected such that the ratio of the left or the right foot in the IGTN and control group was the same.

Their foot posture index-6 components, Staheli's index, radiological hallux valgus angle and active maximum dorsiflexion of the first metatarsophalangeal joint on weight-bearing were measured and compared.

For dependent variables with significant correlation, a one-way multivariate analysis of variance (MANOVA) was carried out to determine if there was a significant difference on the combined dependent variables. For dependent variables without significant correlation, separate independent sample t-tests / welch t-tests were performed.

DETAILED DESCRIPTION:
Precautions were taken to ensure consistency in measurement. To standardize the bisection techniques in measuring radiological hallux valgus angle, this study followed the recommendation from the American Orthopaedic Foot & Ankle Society. The longitudinal axis of the first metatarsal and that of the first proximal phalanx were formed respectively by 2 reference points marked on each of the two bones. The reference points on the first proximal phalanx were 1/2 to 1 cm proximal or distal to the articular surface while the reference points on the first metatarsal were 1 to 2 cm proximal or distal to the articular surface.

The active maximum dorsiflexion of the first metatarsophalangeal joint was measured with goniometer on weight-bearing. The bisection was carried out under a weight-bearing condition to avoid error due to soft-tissue movement when participants changed from a non weight-bearing position to a weight-bearing position.

ELIGIBILITY:
Inclusion criteria for the IGTN group:

* history of ingrown toenails on hallux within 1 year
* dorso-plantar standing view of foot x-ray taken or to be taken

Exclusion criteria for the IGTN group:

* paediatrics (Age<18)
* pincer nails / fungal nails
* prior existence of osteoarticular surgery in the foot
* severe trauma that changes foot morphology
* uncontrolled systemic disease
* pre-existing neurological diseases
* lower limb paralysis or paresis

Inclusion criterion for the control group:

- dorso-plantar standing view of foot x-ray taken or to be taken

Exclusion criteria for the control group:

* all the exclusion criteria of IGTN group
* history of IGTN in his or her lifetime
* flatfoot / first metatarsophalangeal joint pathology as the chief complaint

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients attending the Orthopaedic out-patient clinic at Prince of Wales Hospital in Hong Kong
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2018-04-27 (Actual); Study Completion 2018-04-27 (Actual)

PRIMARY OUTCOMES:
Foot Posture Index-6 components | throughout the study, within 1 year after ingrown toenails for the ingrown toenail group
  * Clinical assessment for flat foot
  * Normal: 0 to +5
  * Pronated: +5 to +9 ; Highly pronated: +10 or above
  * Supinated: -1 to -4; Highly supinated: -5 to -12
Staheli's Index | throughout the study, within 1 year after ingrown toenails for the ingrown toenail group
  * It provides a measurement of flat foot on footprint.
  * The Staheli's index increases as the foot becomes more pronated and is closer to zero as the foot becomes more supinated.
radiological Hallux Valgus Angle | throughout the study, within 1 year after ingrown toenails for the ingrown toenail group
  * Radiological measurement for hallux abducto valgus
  * Normal: <15º
Active maximum dorsiflexion of the first metatarsophalangeal joint on weight bearing | throughout the study, within 1 year after ingrown toenails for the ingrown toenail group
  Clinical measurement with goniometer for hallux limitus

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No